CLINICAL TRIAL: NCT07175038
Title: A Phase 2A, Open-Label Single Arm Multicenter Exploratory Study to Evaluate the Safety, Tolerability, and Efficacy of Oral Doses of ROC-101 in Patients With Pulmonary Arterial Hypertension (PAH) and Pulmonary Hypertension Associated With Interstitial Lung Disease (ILD-PH).
Brief Title: A Study of ROC-101 in Patients With Pulmonary Arterial Hypertension (PAH) and Pulmonary Hypertension Associated With Interstitial Lung Disease (ILD-PH) (ROCSTAR STUDY)
Acronym: ROCSTAR
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AllRock Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROC-101-201
Record Dates: First submitted 2025-09-02; First posted 2025-09-16 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Arterial Hypertension (PAH); Pulmonary Hypertension, Interstitial Lung Disease
Keywords: Rho kinase inhibitor; ROCK inhibitor; Pan ROCK Inhibitor; ROCK-1 and ROCK-2 Inhibitor; ROC-101; PVR; Pulmonary Arterial Hypertension (PAH); Pulmonary Hypertension, Interstitial Lung Disease
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Hypertension, Pulmonary; Lung Diseases, Interstitial; Hereditary Sensory and Autonomic Neuropathies

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ROC-101 Oral Dose (Experimental)
  Interventions: Drug: ROC-101

INTERVENTIONS:
Drug: ROC-101 — Oral, daily administered Rho kinase inhibitor

SUMMARY:
This study evaluates the effect of ROC-101 in adults with either Pulmonary Arterial Hypertension (PAH) or Pulmonary Hypertension Associated with Interstitial Lung Disease (ILD-PH). Each eligible participant will receive standard of care (SOC) plus ROC-101 for a 24-week treatment period, followed by a long-term extension period of the study through the end of the program or marketing approval/authorization.

DETAILED DESCRIPTION:
This is a Phase 2a, open-label, single-arm, multicenter, exploratory study to evaluate the safety, tolerability, and efficacy of oral doses of ROC-101 for the treatment of participants with either World Health Organization (WHO) Group I PAH or WHO Group III ILD-PH.

All eligible PAH/ILD-PH participants will receive SOC therapy plus ROC-101 at a starting dose level of 10 mg orally (PO) daily (QD) and escalating to 40 mg PO QD for the remainder of the main study period of 24 weeks. Evaluations include hemodynamic measures collected during right heart catheterization (RHC) and adverse events.

ELIGIBILITY:
Key Inclusion Criteria:

1. Must be age 18 or older at the time of signing the informed consent form (ICF). The participant must understand and voluntarily sign an ICF prior to any study-related procedures
2. Documented findings on a right heart catheterization (RHC) consistent with a diagnosis World Health Organization (WHO) Group 1 PAH or WHO GROUP 3 PAH
3. Symptomatic Pulmonary Hypertension (PH) classified as WHO Functional Class II or III symptoms
4. PAH participants: Pulmonary Vascular Resistance (PVR) of ≥ 5 Wood units, Pulmonary Capillary Wedge Pressure (PCWP) ≤ 15 mmHg and Mean Pulmonary Arterial Pressure (mPAP) > 20 mm Hg and ILD-PH participants: PVR of ≥ 3 Wood units, PCWP ≤ 15 mmHg and mPAP > 20 mm Hg
5. Participants on stable background therapy for PAH or ILD-PH.
6. Females of childbearing potential (as defined in protocol) must agree to use highly effective contraception (as defined in the protocol)
7. Male participants must follow protocol-specified contraception guidance.
8. Participants must be able to communicate well with Investigators, understand the study procedures in the ICF and are agreeable to complete the study in accordance with the protocol.
9. Must be able to swallow tablets.
10. Pulmonary function tests (PFT):

    PAH participants at Screening as follows:
    1. Forced Vital Capacity (FVC) > 70% predicted; or if between 60% to 70% predicted, or if not possible to be determined, confirmatory High-Resolution Computed Tomography (HRCT) indicating no more than mild (<10% fibrosis) ILD; and
    2. The ratio of FEV1 (first second)/FVC > 0.70 of predicted.

    ILD-PH participants at Screening as follows:
    1. PFTs consistent with their ILD diagnosis and showing FEV1/ FVC ratio > 65% and HRCT > 10% fibrosis, based on the proportion of lung parenchyma affected by fibrotic changes.

       and,
    2. Minimum FVC of 50% and diffusing capacity for carbon monoxide (DLCO) (corrected for Hb g/dl) >25%
11. In PAH participants, i.e., Cohorts 1 and 2 only, ventilation-perfusion (VQ) scan (or, if unavailable, a negative CT pulmonary angiogram [CTPA] or pulmonary angiography result), any time prior to Screening or conducted during the Screening Period, with a normal or low probability result that is not clinically significant
12. Acceptable Electrocardiogram (ECG) findings as assessed by the Investigator or qualified designee at the Screening Visit and at the Baseline Visit (Day 1), including each criterion as listed below:

    * Normal sinus rhythm (HR) between 40 and 100 beats per minute, inclusive);
    * Corrected QT Interval (QTcF) interval ≤ 450 msec (males) and ≤ 460 msec (females);
    * QRS interval ≤ 120 msec; if > 120 msec, result will be confirmed by a manual over read
13. Body weight at the Screening visit and at Baseline (Day 1) is greater than 50.0 kg and the body mass index (BMI) is in the range of 19.00 to 36.00 kg/m2, inclusive
14. 6MWD ≥ 100 and ≤ 550 meters repeated twice, once during Screening Period and once at the Baseline Visit (Day 1) and both values within 15% of each other, allowing for a third repeat if > 15% difference, calculated from the higher/highest value

Key Exclusion Criteria:

1. Diagnosis of PH WHO Groups 2, 4, or 5
2. Diagnosis of the following PAH Group 1 subtypes: human immunodeficiency virus (HIV)-associated PAH, PAH associated with portal hypertension, schistosomiasis-associated PAH and pulmonary veno-occlusive disease and/or pulmonary capillary hemangiomatosis
3. Positive blood test for hepatitis B virus surface antigen (HBsAg), hepatitis C virus (HCV) antibody (HCVAb) (unless participants have had treatment for HCV and have a negative HCV ribonucleic acid [RNA] polymerase chain reaction [PCR]) or HIV antibody
4. Participants with known hypersensitivity to ROC-101 or any components of its formulations
5. History of malignancy within the last 5 years, with the exception of fully excised or treated basal cell carcinoma, cervical carcinoma in-situ, or ≤ 2 squamous cell carcinomas of the skin
6. History of clinically significant (as determined by the Investigator) non-PAH related cardiac, endocrine, hematologic, hepatic, immune, metabolic, urologic, pulmonary, neurologic, neuromuscular, dermatologic, psychiatric, renal, and/or other diseases that may limit participation in the study
7. Participation in another clinical trial involving intervention with another investigational drug, approved therapy for investigational use, or investigational device within 4 weeks prior to Baseline Visit (unless it is in the follow-up period of an interventional study), or if the half-life of the previous product is known, within 5× the half-life prior to Baseline Visit (Day 1), whichever is longer
8. Major surgery within 8 weeks prior to Baseline Visit (Day 1) or major surgery scheduled or planned in the main study. Participants must have completely recovered from any previous surgery prior to the Screening Visit
9. Prior heart or heart-lung transplants, or a participant listed for heart and/or lung transplantation or prior pneumonectomy
10. Pregnant or breastfeeding females
11. Males who do not agree to protocol contraception guidelines
12. Uncontrolled systemic hypertension as evidenced by sitting SBP > 160 mm Hg or sitting diastolic BP > 100 mm Hg during Screening Visit and Baseline Visit (Day 1) after a period of rest
13. Systolic BP < 90 mm Hg during Screening Visit or at Baseline Visit (Day 1)
14. History of known pericardial constriction or a clinically significant (more than trace or trivial [i.e., ≥10 mm]) pericardial effusion seen in diastole or in both systole and diastole on echocardiogram (ECHO) historically and confirmed on screening ECHO
15. RHC contraindicated during the study per Investigator
16. Cerebrovascular accident within 3 months (120 days) of start of Screening
17. History of restrictive or constrictive or congestive cardiomyopathy
18. Left ventricular ejection fraction (LVEF) < 50% on historical echocardiogram (ECHO) performed within 6 months prior to start of Screening period (and confirmed during the Screening ECHO) or grade 2 or higher diastolic dysfunction
19. Any current symptomatic coronary disease (myocardial infarction, percutaneous coronary intervention, coronary artery bypass graft surgery, or cardiac anginal chest pain in the past 6 months (180 days) prior to start of Screening)
20. History of acutely decompensated left heart failure or right heart failure within 90 days prior to Baseline, as per Investigator assessment
21. Significant (≥ 2+ [or > mild] regurgitation) mitral regurgitation or aortic regurgitation valvular disease, or more than mild mitral stenosis or aortic stenosis valvular disease as seen on Screening ECHO
22. Started or stopped receiving any general supportive therapy for PH (e.g., oxygen, anticoagulants, digoxin) within 30 days prior to start of Screening
23. Use of supplemental oxygen > 10 liters/minute and SaO2 < 90% while receiving typical oxygen supplementation
24. Received intravenous (IV) inotropes (e.g., dobutamine, dopamine, norepinephrine, vasopressin) within 30 days prior to start of Screening
25. History of atrial septostomy within 180 days prior to start of Screening
26. History of portal hypertension or chronic liver disease, defined as mild to severe hepatic impairment (Child-Pugh Classes A to C)
27. Untreated, severe (defined as apnea hypoxia index of > 30) obstructive sleep apnea
28. Active daily smoker of cannabis or tobacco
29. Current alcohol abuse or current illicit drug use
30. WHO Group 3 due to severe chronic obstructive pulmonary disease (COPD) or chronic pulmonary fibrosis and emphysema (CPFE) or PFT with FVC < 50% or FEV1/FVC < 65% or DLCO < 25% (corrected for Hb g/dl)
31. Presence of lab abnormalities at Screening
32. History of greater than severe renal disease, including any episode of acute renal failure, with or without a prior history of renal disease in which acute dialysis (e.g., intermittent hemodialysis or continuous veno-venous hemofiltration) was required
33. Initiation of an exercise program for cardiopulmonary rehabilitation within 90 days prior to Baseline or planned initiation during the study (participants who are stable in the maintenance phase of a program and who will continue for the duration of the study are eligible)
34. Participants who plan to continue, or start during the study, medications which are sensitive cytochrome (CYP) 2D6 substrates with a narrow therapeutic index, such as nortriptyline, venlafaxine, and amitriptyline or CYP1A2 substrates with a narrow therapeutic index
35. History or presence of impaired cardiac function
36. Participants who plan to donate blood after signing consent for the study and for 28 days after their last dose of study drug

Key Inclusion Criteria for Extension Period:

1. Participants must complete the main study period (defined as completion of assessments through the Week 24 visit)
2. Women of child-bearing potential (WOCBP) must have negative pregnancy test
3. All participants must comply with contraceptive guidance until 28 days after last dose of study drug for WOCBP and 90 days after the last dose of study drug for males

Key Exclusion Criteria for Extension Period:

1. Participant withdrew from main study period due to an AE related to study drug
2. Female participant who is pregnant, breastfeeding, or intends to conceive during the long-term extension period
3. Males who do not agree to follow protocol contraception guidelines
4. Any condition that in the opinion of the investigator may pose a risk to the participant, interferes with the participant's participation or confounds assessments of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Change in Pulmonary Vascular Resistance (PVR) from Baseline versus at 24 weeks | Baseline and 24 weeks
  Each participant's PVR, at resting supine, was measured by Right Heart Catheterization (RHC) at baseline and at 24 weeks.
Safety assessments: Number of Participants Who Experienced an Adverse Event (AE) | 24 Weeks
  Number of Participants Who Experienced an Adverse Event (AE)

SECONDARY OUTCOMES:
Change in 6-minute Walk Distance (6MWD) from Baseline versus at 24 weeks | Baseline and 24 Weeks
  The 6MWD was the distance walked in 6 minutes as a measure of functional capacity. This was assessed using the 6-minute walk test (6MWT). Per protocol, change from baseline in 6MWD at Week 24 will be measured
Change in NT-proBNP from Baseline versus at 24 weeks | Baseline and 24 Weeks
  NT-proBNP is a circulating biomarker that reflects myocardial stretch and is one of the biomarkers measured. The change from baseline in NT-proBNP level versus at Week 24 will be measured.
Change in World Health Organization (WHO) Functional Classification | Baseline and 24 weeks
  The severity of participant's pulmonary arterial hypertension (PAH) symptoms will be graded using the WHO FC system. WHO functional classification for PAH ranges from Class I (no limitation in physical activity, no dyspnea with normal activity), Class II (slight limitation of physical activity), Class III (marked limitation of physical activity) and Class IV (cannot perform a physical activity without any symptoms, dyspnea at rest). Participants who improve in WHO FC were classified into "Improved", "No change" and "Worsened". Improvement = reduction in FC, worsened = increase in FC and no change = no change in FC. Percentage of participants who improve in WHO FC at Week 24 from baseline will be reported.
Change in Right Atrial Pressure (RAP) measured by Right Heart Catheterization (RHC) | Baseline and 24 weeks
Change in Mean Pulmonary Artery Pressure (mPAP) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Change in Cardiac Output (CO) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Change in Cardiac Index (CI) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Change in Pulmonary Capillary Wedge Pressure (PCWP) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Changes in Mixed Venous Oxygen Saturation (SvO2) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Changes in Stroke Volume (SV) SV index (SVI) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Change in Pulse Pressure (PP) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks
Changes in Pulmonary Artery Compliance (PAC) measured by Right Heart Catheterization (RHC) | Baseline and 24 Weeks

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Mayo Clinic of Florida, Jacksonville, Florida
  - The University of Kansas Medical Center Research Institute, Kansas City, Kansas
  - Bend Memorial Clinic, Bend, Oregon

IPD SHARING:
Plan to Share IPD: No